CLINICAL TRIAL: NCT05607043
Title: Rutgers Pilot for Pragmatic Return to Effective Dental Infection Control Through Triage and Testing (PREDICT)- Patient LAB Test
Brief Title: Rutgers Pilot for PREDICT- Patient LAB Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Cecile A. Feldman, DMD, Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro2020002999; X01DE030407 (Other: NIDCR)
Record Dates: First submitted 2022-10-31; First posted 2022-11-07 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: SARS-CoV2 Infection
Keywords: Screening; Lab-based testing; Asymptomatic patients; Perception of safety; Feasibility
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Pilot study to assess feasibility of testing asymptomatic dental patients for SARS-CoV-2 antigen using lab-based RNA RT-PCR testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- SARS-CoV-2 testing (Other): There is only one arm in this study- the study is a non-randomized pilot. All the subjects will be tested for SARS CoV 2 viral infection as described.
  Interventions: Device: Testing for SARS CoV2 RNA

INTERVENTIONS:
Device: Testing for SARS CoV2 RNA — Device: Testing for SARS CoV2 RNA- lab-based RNA RT-PCR testing

SUMMARY:
A pilot study was initiated to assess feasibility of testing asymptomatic dental patients presenting to the Oral Medicine Clinic at Rutgers School of Dental Medicine for SARS-CoV-2 viral RNA using an FDA approved RT-PCR test for SARS-CoV2- an RNA RT-PCR assay (Accurate Diagnostics)

DETAILED DESCRIPTION:
Patients with upcoming dental appointments at the Oral Medicine clinic at Rutgers School of Dental Medicine were contacted to solicit interest in participating in a pilot study to assess feasibility of testing asymptomatic dental patients for SARS CoV 2 infection using an RNA RT-PCR assay. Interested subjects completed a previsit survey after confirming their interest electronically. Subsequently, they received kit to collect their saliva sample at home along with instructions on how to do so. They were directed to drop off their saliva samples for testing at the dental clinic and signed the consent form at that time. After confirming a negative result, the patients were subsequently triaged over the phone for any symptoms and the following day, presented for their dental visit.

On the day of their visit, they were triaged, completed their dental visit and were surveyed to get their feedback on the study procedures and their perceptions of safety.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years or older; reporting to the Rutgers School of Dental Medicine for a dental visit

Exclusion Criteria:

* Previous participation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-01-31 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cecile A Feldman, Principal Investigator — Rutgers School of Dental Medicine
Locations (1):
- Rutgers School of Dental Medicine, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
If the COVID test results show that a participant is positive for COVID-19, the study staff will tell the participant the results. The study staff will be required to give the participant's name to the state's Department of Public Health if the participant tests positive because this is the law.
  At the end of the study, de-identified data will be provided to the National Coordinating Center.

REFERENCES:
- [Background] American Dental Association COVID-19 Toolkit - Update to Office Procedures During COVID-19. https://www.ada.org/-/media/project/ada-organization/ada/ada-org/files/resources/coronavirus/update_to_office_procedures_during_covid19.pdf accessed on November 11, 2021.
- [Background] Estrich CG, Mikkelsen M, Morrissey R, Geisinger ML, Ioannidou E, Vujicic M, Araujo MWB. Estimating COVID-19 prevalence and infection control practices among US dentists. J Am Dent Assoc. 2020 Nov;151(11):815-824. doi: 10.1016/j.adaj.2020.09.005. PMID 33071007
- [Background] Shirazi S, Stanford CM, Cooper LF. Testing for COVID-19 in dental offices: Mechanism of action, application, and interpretation of laboratory and point-of-care screening tests. J Am Dent Assoc. 2021 Jul;152(7):514-525.e8. doi: 10.1016/j.adaj.2021.04.019. Epub 2021 May 4. PMID 34176567

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 11 asymptomatic dental patients with upcoming appointments at the Oral Medicine clinic, Rutgers School of Dental Medicine, were enrolled. Study participation ranged from January- February 2021.
Period: Overall Study
Arm/Group | SARS-CoV-2 Testing
Started | 11
Completed | 9
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | SARS-CoV-2 Testing
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (7.651)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 0
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Patient Willingness to Participate in the Study
Description: Percentage of 36 patients who were approached to enroll in the study who actually enrolled
Time Frame: Day 1
Population: 36 patients were approached to enroll in the study. The percentage of 36 patients who consented to participate in the study is tabulated
Measure: Number; unit: percentage
Arm/Group | SARS-CoV-2 Testing
Number analyzed (Participants) | 36
percentage | 30

2. Primary Outcome: Willingness/Ability to Follow Through With the Study With Surveys, Triage and Testing
Description: Percentage of patients who complete the study
Time Frame: 26 days
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 Testing
Number analyzed (Participants) | 11
Participants | 9

3. Primary Outcome: Patient Test Completion
Description: Percentage of patients with completed SARS-CoV-2 testing
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 Testing
Number analyzed (Participants) | 11
Participants | 10

4. Primary Outcome: Percentage of Subjects Who Complete Study Activities to Optimize Gap Between Testing and Study Visit
Description: Percentage of subjects completing study activities within the defined optimal window
Time Frame: From initial consent through study completion- approximately 4 weeks
Measure: Number; unit: participants
Arm/Group | SARS-CoV-2 Testing
Number analyzed (Participants) | 11
participants | 9

5. Primary Outcome: Ease of Complying With Protocol
Description: Number of participants indicating that it was easy to complete the surveys
Time Frame: Day 26
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 Testing
Number analyzed (Participants) | 11
Participants | 8

6. Primary Outcome: Percent of Patients Who Completed All of the Required Surveys
Description: Percentage of patients participating in the study who completed pre-visit, triage and post-visit surveys
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 Testing
Number analyzed (Participants) | 11
Participants | 9

ADVERSE EVENTS:
Time Frame: From signing initial consent to completion of study visit- approximately 4 weeks
Description: This study involved a nasal swab, and a survey
Arm/Group | SARS-CoV-2 Testing
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/43/NCT05607043/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/43/NCT05607043/ICF_001.pdf